CLINICAL TRIAL: NCT04618744
Title: A Double-Blind, Randomized, Placebo-controlled, Multi-center Study to Assess the Safety and Efficacy of Oral Insulin to Reduce Liver Fat Content in Type 2 Diabetes Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Study to Assess the Safety and Efficacy of Oral Insulin in T2DM Patients With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA-D-N02
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2; NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — ORMD-0801; Insulin; Capsules; Fish Oils

STUDY DESIGN:
Intervention Model Description: The study will consist of a Screening Phase, Placebo Run-in Phase, Treatment Phase, and an End-of-Study Phase. Approximately 36 subjects will be randomized in a 2:1 ratio to receive either 8 mg ORMD-0801, 1 capsule twice a day (once in the morning approximately 30 to 45 minutes prior to breakfast and no later than 10 AM, and once at night between 8 PM to Midnight and no sooner than 1 hour after dinner) or matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Fish oil
  Interventions: Other: Placebo
- ORMD-0801 (Insulin) capsule 8 mg BD (Experimental): ORMD-0801 (insulin) capsule Dose: 8 mg BD Dosage Regimen: 1 capsule twice a day (once in the morning approximately 30 to 45 minutes prior to breakfast and no later than 10 AM, and once at night between 8 PM to Midnight and no sooner than 1 hour after dinner) Mode of Administration: Oral
  Interventions: Drug: ORMD-0801 (Insulin) capsule 8 mg BD

INTERVENTIONS:
Drug: ORMD-0801 (Insulin) capsule 8 mg BD — 8 mg ORMD-0801, 1 capsule, twice a day, once in the morning and once in the evening.
  Other Names: Oral Insulin
  Arms: ORMD-0801 (Insulin) capsule 8 mg BD
Other: Placebo — Matching Placebo
  Other Names: Fish oil
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, multi-center study using the oral ORMD-0801 insulin formulation in patients with NASH and confirmed type 2 DM.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, multi-center study using the oral ORMD-0801 insulin formulation in patients with NASH and confirmed type 2 DM. The study will consist of a Screening Phase, Placebo Run-in Phase, Treatment Phase and an End-of-Study Phase. Approximately 36 subjects will be randomized in a 2:1 ratio to receive either 8 mg ORMD-0801, 1 capsule twice a day (once in the morning approximately 30 to 45 minutes prior to breakfast and no later than 10 AM, and once at night between 8 PM to Midnight and no sooner than 1 hour after dinner) or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-70 years.
* BMI ≥25
* Known type 2 DM according to American Diabetic Association (one of the three needed): Fasting Plasma Glucose ≥126 mg/dl or 2h postprandial (PG) following 75g OGTT ≥200 mg/dl or HbA1c > 6.5%28 or on treatment with metformin only or metformin in addition to no more than two of the following medications sulfonylurea, DPP-4 inhibitors, GLP-1 receptor agonists, Thiazolidinediones (TZDs)
* Diagnosis of NAFLD by non-invasive determination of hepatic steatosis grade S1, defined as hepatic steatosis>8% by MRI- PDFF and CAP FibroScan ≥ 238 dB/m.
* Liver enzyme abnormalities: ULN≤5 times.
* Fibrosis score 21≤F≤3 as defined by FibroScan measurement (Liver stiffness measurement, LSM) of 6 ≤ LSM ≤ 12 kPa.
* Signature of the written informed consent.
* Negative urine serum pregnancy test at Screening study entry for females of childbearing potential (WCBP).
* WCBP must have a negative urine pregnancy test result prior to the start of the run-in period and initiation if active dosing. A negative urine and serum pregnancy test must be obtained prior to active dosing. Males and females of childbearing potential must use two methods of contraception (double barrier method), one of which must be an acceptable barrier method from the time of screening to the last dosing study visit (22 weeks). Barrier methods of contraception include male condoms plus spermicide, diaphragm with spermicide plus male condom, cervical cap with spermicide plus male condom, or oral contraceptives. Acceptable methods of birth control include abstinence, oral contraceptives, surgical sterilization, vasectomy, the contraceptive patch, and the contraceptive ring. If a subject is not usually sexually active but becomes active, he or his partner should use medically accepted forms of contraception. Sperm donations will not be allowed for the duration of the study and for 90 days after the last dose of study drug.
* Females of non-childbearing potential are defined as postmenopausal who a) had more than 24 months since last menstrual cycle with menopausal levels of FSH (FSH Level > 40), b) who are surgically menopausal (surgical sterility defined by tubal occlusion, bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* For hypertensive patients, hypertension must be controlled by a stable dose of anti-hypertensive medication for at least 2 months prior to screening (and the stable dose can be maintained throughout the study) with BP < 150/<95 mmHg
* Patients previously treated with vitamin E (>400IU/day), Polyunsaturated fatty acid (>2g/day) or Ursodeoxycholic acid fish oil can be included if drugs are stopped at least 3 months prior to enrolment and up to the end of the study.
* Glycaemia must be controlled (Glycosylated Hemoglobin A1C ≤8.5%) while any HbA1C increment should not exceed 1% during 6 months prior to enrolment).

Exclusion Criteria:

* Patients with active (acute or chronic) liver disease other than NASH (e.g. viral hepatitis, genetic hemochromatosis, Wilson disease, alpha-1 antitrypsin deficiency, alcohol liver disease, drug-induced liver disease) at the time of enrolment.
* ALT or AST > 5 times ULN.
* Abnormal synthetic liver function (serum albumin ≤3.5gm%, INR >1.3).
* Known alcohol and/or any other drug abuse or dependence in the last five years.
* Weight >120 Kg (264.6 lbs.)
* Known history or presence of clinically significant, cardiovascular, gastrointestinal, metabolic (other than diabetes mellitus), neurologic, pulmonary, endocrine, psychiatric, neoplastic disorder, or nephrotic syndrome.
* History or presence of any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolites (e.g. inflammatory bowel disease (IBD), previous intestinal (ileal or colonic) operation, chronic pancreatitis, celiac disease, or previous vagotomy.
* Weight loss of more than 5% within 6 months prior to enrolment.
* History of bariatric surgery.
* Uncontrolled blood pressure BP ≥150/≥95.
* Non-type 2 DM (type 1, endocrinopathy, genetic syndromes etc.).
* Patients with HIV.
* Daily alcohol intake >20 g/day (2 units/day) for women and >30 g/day (3 units/day) for men.
* Treatment with anti-diabetic medications other than metformin and more than two of the following medications sulfonylurea, DPP-4 inhibitors, GLP-1 receptor agonists, TZDs
* Metformin, fibrates, statins, not provided on a stable dose in the last 6 months.
* Patients who are treated with valproic acid, Tamoxifen, methotrexate, amiodarone.
* Chronic treatment with antibiotics (e.g. Rifaximin).
* Homeopathic and/or Alternative treatments. Any treatment must be stopped before the screening period.
* Uncontrolled hypothyroidism defined as Thyroid Stimulating Hormone >2X the upper limit of normal (ULN). Thyroid dysfunction controlled for at least 6 months prior to screening is permitted.
* Patients with renal dysfunction: eGFR< 40 ml/min.
* Unexplained serum creatinine phosphokinase (CPK) >3X the upper limit of normal (ULN). Patients with a reason for CPK elevation may have the measurement repeated prior to enrolment; a CPK retest > 3X ULN leads to exclusion.
* Subjects meeting criteria for contraindication for MRI - including the following:

  i. History of severe claustrophobia impacting the ability to perform MRI during the study, even despite mild sedation/treatment with as anxiolytic.

ii. Subjects with metal implants, devices, paramagnetic objects contained within the body, and excessive or metal-containing tattoos.

iii. Subjects unable to lie still within the environment of the MRI scanner or maintain a breath-hold for the required period to acquire images, even despite mild sedation/treatment with an anxiolytic.

* The subject participated in a clinical research study involving a new chemical entity within 4 weeks of study entry.
* Known allergy to soy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kidron, Ph.D., Study Director — Oramed, Ltd.; Joel M Neutel, M. D., Principal Investigator — Integrium
Locations (3):
- Orange County Research Center, Tustin, California, United States
- Israel (2):
  - Hadassah Medical Center, Jerusalem, International/Other
  - Tel Aviv Sourasky Medical Center- Ichilov Hospital, Tel Aviv, International/Other

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin SC, Heba E, Bettencourt R, Lin GY, Valasek MA, Lunde O, Hamilton G, Sirlin CB, Loomba R. Assessment of treatment response in non-alcoholic steatohepatitis using advanced magnetic resonance imaging. Aliment Pharmacol Ther. 2017 Mar;45(6):844-854. doi: 10.1111/apt.13951. Epub 2017 Jan 24. PMID 28116801
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Ratziu V, Bellentani S, Cortez-Pinto H, Day C, Marchesini G. A position statement on NAFLD/NASH based on the EASL 2009 special conference. J Hepatol. 2010 Aug;53(2):372-84. doi: 10.1016/j.jhep.2010.04.008. Epub 2010 May 7. No abstract available. PMID 20494470
- [Background] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Background] Germain T, Favelier S, Cercueil JP, Denys A, Krause D, Guiu B. Liver segmentation: practical tips. Diagn Interv Imaging. 2014 Nov;95(11):1003-16. doi: 10.1016/j.diii.2013.11.004. Epub 2013 Dec 30. PMID 24388431
- [Derived] Ishay Y, Neutel J, Kolben Y, Gelman R, Arbib OS, Lopez O, Katchman H, Mohseni R, Kidron M, Ilan Y. Oral Insulin Alleviates Liver Fibrosis and Reduces Liver Steatosis in Patients With Metabolic Dysfunction-associated Steatohepatitis and Type 2 Diabetes: Results of Phase II Randomized, Placebo-controlled Feasibility Clinical Trial. Gastro Hep Adv. 2023 Dec 7;3(3):417-425. doi: 10.1016/j.gastha.2023.11.016. eCollection 2024. PMID 39131144

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All screened participants must have an MRI scan prior to enrollment to confirm satisfying the entry criteria of MR PDFF >= 8%
Period: Overall Study
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Started | 11 | 21
Completed | 11 | 19
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD | Total
Number analyzed (Participants) | 11 | 21 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.73 (10.355) | 58.67 (7.565) | 58.00 (8.508)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 6 | 14 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 18
  Not Hispanic or Latino | 4 | 10 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 19 | 29
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 32.109 (4.5496) | 33.567 (5.2981) | 33.066 (5.0281)
Childbearing Status [Count of Participants; unit: Participants]
  Of Childbearing Potential | 0 | 0 | 0
  Surgically Sterilized | 2 | 4 | 6
  At least 24 months Post-Menopausal | 3 | 3 | 6
  Not Applicable | 6 | 14 | 20
Median Magnetic Resonance Proton Fat Fraction (MRPDFF) [Median (Full Range); unit: percent liver fat] — Median Magnetic Resonance Proton Density Fat Fraction (MRPDFF) of Liver Segment 3, according to the Couinaud classification of hepatic segments.
  percent liver fat | 21.100 [6.97 to 33.50] | 13.900 [5.34 to 26.90] | 14.250 [5.34 to 33.50]

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events
Description: The Number of Treatment-Emergent Adverse Events (TEAE) according to CTCAE version 4.03. A TEAE is an adverse event for which the start date is on or after the date that the treatment began.
Time Frame: Screening through Week 16
Population: Safety Population
Measure: Number; unit: Adverse Events
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
Adverse Events | 0 | 2

2. Secondary Outcome: Median MRPDFF at Baseline and Week 12 of Whole Liver
Description: Median MRPDFF at Baseline and Week 12 of Whole Liver. Delineation by a central radiologist of the whole liver in the slice with the largest liver cross-section. The Liver was subdivided into 8 sections according to the Coinaud liver segmentation for MRI.
Time Frame: Baseline and Week 12 (Visit 8)
Population: Intent-to-Treat. Placebo population: One subject's baseline Whole Liver MRPDFF was missing. This patient did have their Visit 8 MRI, however since there was no baseline MRPDFF Whole Liver, the change from baseline measurement cannot be calculated. A second patient did not have their Visit 8 MRI acquired.
  ORMD-0801:One subject did not have a Visit 8 MRI (discontinued study due to Withdrew Consent). A second subject did not have a Visit 8 MRI (discontinued study due to Adverse Event)
Measure: Median (Full Range); unit: Percent fat (MRPDFF)
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
Percent fat (MRPDFF)
  Median MRPDFF at Baseline: number analyzed (Participants) | 10 | 21
  Median MRPDFF at Baseline | 24.350 [9.80 to 31.90] | 15.340 [5.34 to 27.20]
  Median MRPDFF (percentage fat) at Week 12: number analyzed (Participants) | 10 | 19
  Median MRPDFF (percentage fat) at Week 12 | 17.300 [3.66 to 29.50] | 13.300 [3.33 to 26.80]

3. Secondary Outcome: Percent Change From Baseline of Median MRPDFF of Whole Liver
Description: The percent change in MR PDFF from baseline to Week 12 of Whole Liver
Time Frame: Baseline and Week 12 (Visit 8)
Population: Intent-to-Treat. Placebo population: One subject's baseline Whole Liver MRPDFF was missing. This patient did have their Visit 8 MRI, however since there was no baseline MRPDFF Whole Liver, the change from baseline measurement cannot be calculated. A second patient did not have their Week 12 MRI acquired.
  ORMD-0801:One subject did not have a Visit 8 MRI (discontinued study due to Withdrew Consent). A second subject did not have a Visit 8 MRI (discontinued study due to Adverse Event)
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 9 | 19
percent change | -1.103 [-28.97 to 16.33] | -7.105 [-65.78 to 59.18]

4. Secondary Outcome: Mean Magnetic Resonance Proton Density Fat Fraction (MRPDFF) of Whole Liver
Description: Mean Magnetic Resonance Proton Density Fat Fraction (MRPDFF) of Whole Liver at Baseline and Week12. The Whole liver was delineated by a central radiologist. The liver was subdivided into 8 sections according to the Coinaud liver segmentation for MRI.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 10 | 21
percentage of fat
  Mean MRPDFF of Whole Liver at Baseline | 21.558 (8.2072) | 15.683 (6.1605)
  Mean MR PDFF of Whole Liver at Week 12: number analyzed (Participants) | 10 | 19
  Mean MR PDFF of Whole Liver at Week 12 | 17.414 (8.6331) | 14.274 (6.8032)

5. Secondary Outcome: Percent Change From Baseline in Mean Magnetic Resonance Proton Density Fat Fraction (MRPDFF) of Whole Liver
Description: The percent change from basline in liver fat content as measured by the mean MRI Proton density Fat Fraction (MR PDFF) at baseline and at week 12 of Whole Liver
Time Frame: Screening and Week 12 (Visit 8)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of change in MRPDFF
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 9 | 19
Percentage of change in MRPDFF | -6.526 (15.3158) | -7.489 (27.3972)

6. Secondary Outcome: Median Magnetic Resonance Proton Density Fat Fraction (MR PDFF) of Liver Segment 3
Description: Median MRPDFF (percentage fat in the liver) of liver segment 3 as measured by MRI Proton Density Fat Fraction at baseline and at week 12. Delineation by a central radiologist of the Liver Segment 3 in the slice with the largest Liver Segment 3 cross-section.
Time Frame: Baseline and Week 12 (Visit 8)
Population: Intent-to-Treat. Placebo population: One subject's baseline Liver Segment 3 radius was missing. This patient did have their Visit 8 MRI, however since there was baseline data missing, the change from baseline measurement cannot be calculated. A second patient did not have their Week 12 MRI acquired.
  ORMD-0801:One subject did not have a Visit 8 MRI (discontinued study due to Withdrew Consent). A second subject did not have a Visit 8 MRI (discontinued study due to Adverse Event)
Measure: Median (Full Range); unit: percentage fat
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
percentage fat
  Median MRPDFF Liver Segment 3 Baseline | 21.10 [6.97 to 33.50] | 13.900 [5.34 to 26.90]
  Median MRPDFF Liver Segment 3 Week 12: number analyzed (Participants) | 10 | 19
  Median MRPDFF Liver Segment 3 Week 12 | 15.150 [3.11 to 28.70] | 11.900 [3.28 to 26.43]

7. Secondary Outcome: Percent Change From Baseline of Median MRPDFF of Liver Segment 3
Description: Percent Change from Baseline Median MRPDFF of Liver Segment measured at baseline and Week 12 (Visit 8)
Time Frame: Baseline and Week 12 (Visit 8)
Population: ntent-to-Treat. Placebo population: One subject's baseline Liver Segment 3 radius was missing. This patient did have their Visit 8 MRI, however since there was baseline data missing, the change from baseline measurement cannot be calculated. A second patient did not have their Week 12 MRI acquired.
  ORMD-0801:One subject did not have a Visit 8 MRI (discontinued study due to Withdrew Consent). A second subject did not have a Visit 8 MRI (discontinued study due to Adverse Event)
Measure: Median (Full Range); unit: percentage change
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 9 | 19
percentage change | 0.000 [-26.97 to 26.40] | -6.424 [-66.67 to 10.19]

8. Secondary Outcome: Mean MRPDFF of Liver Segment 3
Description: Mean MRPDFF of Liver Segment measured at baseline and Week 12
Time Frame: Baseline and Week 12 (Visit 8)
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: percentage fat
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
percentage fat
  MRPDFF of Liver Segment 3 at baseline | 20.617 (9.1032) | 14.560 (5.3974)
  MR PDFF of Liver Segment 3 at Week 12: number analyzed (Participants) | 10 | 19
  MR PDFF of Liver Segment 3 at Week 12 | 16.610 (9.2736) | 13.119 (6.2239)

9. Secondary Outcome: Percent Change of Mean MRPDFF of Liver Segment 3
Description: Percent change from baseline of mean MR PDFF measurement of liver segment 3 at baseline and week 12
Time Frame: Baseline and Week 12 (Visit 8)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of Change in MR PDFF
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 9 | 19
percentage of Change in MR PDFF | 0.105 (17.2630) | -10.763 (20.9231)

10. Secondary Outcome: Median MR PDFF of Liver Segment 6
Description: Median Magnetic Resonance Proton Density Fat Fraction of Liver Segment 6 measured at baseline and at week 12 (Visit 8). Delineation by a central radiologist of Liver Segment 6 in the slice with the largest Liver Segment 6 cross-section.
Time Frame: Screening and Week 12 (Visit 8)
Population: Intent-to-Treat. Placebo population: One subject's baseline Liver Segment 6 radius was missing. This patient did have their Visit 8 MRI, however since there was baseline data missing, the change from baseline measurement cannot be calculated. A second patient did not have their Week 12 MRI acquired.
  ORMD-0801:One subject did not have a Visit 8 MRI (discontinued study due to Withdrew Consent). A second subject did not have a Visit 8 MRI (discontinued study due to Adverse Event)
Measure: Median (Full Range); unit: percentage of liver fat
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
percentage of liver fat
  Median MRPDFF of Liver Segment 6 Baseline | 22.900 [8.76 to 37.00] | 15.420 [4.81 to 30.00]
  Median MRPDFF of Liver Segment 6 Week 12: number analyzed (Participants) | 10 | 19
  Median MRPDFF of Liver Segment 6 Week 12 | 15.400 [3.28 to 27.40] | 12.600 [5.19 to 27.13]

11. Secondary Outcome: Percent Change From Baseline of Median MR PDFF of Liver Segment 6
Description: Percent Change from Baseline of Median Magnetic Resonance Proton Density Fat Fraction of Liver Segment 6 measured at baseline and at week 12
Time Frame: Screening and Week 12 (Visit 8)
Population: as for outcome 10
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 9 | 19
percent change | -4.965 [-37.19 to 15.01] | -6.488 [-41.49 to 54.63]

12. Secondary Outcome: Mean MR PDFF of Liver Segment 6
Description: Mean Magnetic Resonance Proton Density Fat Fraction of Liver Segment 6 measured at baseline and at week 12 (Visit 8)
Time Frame: Screening and Week 12 (Visit 8)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage liver fat
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
percentage liver fat
  Mean MRPDFF of liver segment 6 at Baseline | 22.174 (8.9629) | 15.828 (7.3523)
  Mean MRPDFF of Liver segment 6 at Week 12: number analyzed (Participants) | 10 | 21
  Mean MRPDFF of Liver segment 6 at Week 12 | 16.226 (8.4452) | 14.009 (7.1855)

13. Secondary Outcome: Percent Change From Baseline of Mean MR PDFF of Liver Segment 6
Description: Percent Change from Baseline Mean Magnetic Resonance Proton Density Fat Fraction of Liver Segment 6 measured at baseline and at week 12 (Visit 8)
Time Frame: Screening and Week 12 (Visit 8)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 9 | 19
percent change | -9.891 (15.3865) | -9.310 (21.7602)

14. Secondary Outcome: Median MRPDFF of Liver Segment 8
Description: Median MRPDFF of Liver Segment 8 measured at baseline and Week 12 (Visit 8)
Time Frame: Baseline and Week 12 (Visit 8)
Population: Intent-to-Treat. Placebo population: One subject's baseline Liver Segment 8 radius was missing. This patient did have their Visit 8 MRI, however since there was baseline data missing, the change from baseline measurement cannot be calculated. A second patient did not have their Week 12 MRI acquired.
  ORMD-0801:One subject did not have a Visit 8 MRI (discontinued study due to Withdrew Consent). A second subject did not have a Visit 8 MRI (discontinued study due to Adverse Event)
Measure: Median (Full Range); unit: percentage liver fat
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
percentage liver fat
  Median MRPDFF of Liver Segment 8 at baseline | 25.100 [8.06 to 31.20] | 15.600 [6.63 to 28.20]
  Median MR PDFF of Liver Segment 8 at Week 12: number analyzed (Participants) | 10 | 19
  Median MR PDFF of Liver Segment 8 at Week 12 | 18.200 [3.66 to 27.90] | 13.500 [3.27 to 28.03]

15. Secondary Outcome: Percent Change in Median MRPDFF of Liver Segment 8
Description: Percent change from baseline in median MRPDFF of Liver segment 8 measured at baseline and week 12 (Visit 8).
Time Frame: Baseline and Week 12 (Visit 8)
Population: as for outcome 14
Measure: Median (Full Range); unit: percent change of the median MRPDFF
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 9 | 19
percent change of the median MRPDFF | -6.376 [-35.71 to 12.54] | -5.419 [-65.18 to 32.75]

16. Secondary Outcome: Mean MRPDFF of Liver Segment 8
Description: Liver fat percentage of liver segment 8 as measured by MRI Proton Density Fat Fraction (MR PDFF) at baseline and at week 12 (Visit 8). Delineation by a central radiologist of Liver Segment 8 in the slice with the largest Liver Segment 8 cross-section.
Time Frame: Baseline and Week 12 (Visit 8)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percentage fat
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
percentage fat
  Mean MRPDFF of liver segment 8 at Baseline | 22.565 (7.8978) | 16.071 (6.3147)
  Mean MRPDFF of Liver segment 8 at Week 12: number analyzed (Participants) | 10 | 19
  Mean MRPDFF of Liver segment 8 at Week 12 | 17.451 (2.8338) | 14.817 (7.1945)

17. Secondary Outcome: Percent Change From Baseline in Mean MRPDFF of Liver Segment 8
Description: Percent change from baseline in MRPDFF of liver segment 8 at baseline and at week 12 (Visit 8)
Time Frame: Baseline and Week 12 (Visit 8)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percentage change in MRPDFF
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 9 | 19
percentage change in MRPDFF | 17.451 (8.6343) | 14.817 (7.1945)

18. Secondary Outcome: Liver Steatosis
Description: Liver steatosis measured by FibroScan® at baseline and at week 12 (Visit 8), in units of decibels per meter (dB/M)
Time Frame: Baseline and Week 12 (Visit 8)
Population: Safety Population
Measure: Median (Inter-Quartile Range); unit: dB/M
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
dB/M
  Median Liver Steatosis Baseline | 335 [276 to 345] | 329 [299 to 357]
  Median Liver Steatosis Week 12: number analyzed (Participants) | 11 | 19
  Median Liver Steatosis Week 12 | 345.0 [320.0 to 360.0] | 329.0 [279.0 to 351.0]

19. Secondary Outcome: Change in Liver Steatosis From Baseline
Description: Change in Liver steatosis from baseline measured by FibroScan® at baseline and at week 12 (Visit 8), in units of decibels per meter (dB/M)
Time Frame: Baseline and Week 12 (Visit 8)
Population: Safety Population. One subject did not have a Visit 8 Fibroscan (discontinued study due to Withdrew Consent)
  A second subject did not have a Visit 8 Fibroscan (discontinued study due to Adverse Event)
Measure: Median (Inter-Quartile Range); unit: dB/M
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 19
dB/M | 13.0 [0.0 to 38.0] | -16.0 [-38.0 to 22]

20. Secondary Outcome: Liver Fibrosis
Description: Liver fibrosis measured by FibroScan® at baseline and at week 12 (Visit 8), in units of kilo Pascals (kPa).
Time Frame: Baseline and Week 12 (Visit 8)
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: kPa (kilo Pascals)
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 21
kPa (kilo Pascals)
  Median Liver Fibrosis Baseline | 8.4 [6.4 to 9.0] | 8.6 [6.7 to 9.2]
  Median Liver Fibrosis Week 12: number analyzed (Participants) | 11 | 19
  Median Liver Fibrosis Week 12 | 7.4 [6.5 to 8.7] | 7.4 [6.4 to 9.7]

21. Secondary Outcome: Change From Baseline of Liver Fibrosis
Description: The change from baseline in liver fibrosis measured by FibroScan® at baseline and at week 12 (Visit 8), in units of kilo Pascals (kPa).
Time Frame: Baseline and Week 12 (Visit 8)
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: kPa (kilo Pascals)
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
Number analyzed (Participants) | 11 | 19
kPa (kilo Pascals) | 0.3 [-2.6 to 2.3] | -0.8 [-2.5 to 3.8]

ADVERSE EVENTS:
Time Frame: Placebo Run-In (Week -2) through End-of-Study (Week 16); total of 18 weeks.
Description: NCI CTCAE v. 4.03
Arm/Group | Placebo | ORMD-0801 (Insulin) Capsule 8 mg BD
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/21
Other Adverse Events (participants affected / at risk) | 4/11 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | ORMD-0801 (Insulin) Capsule 8 mg BD (N=21)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointenstinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | ORMD-0801 (Insulin) Capsule 8 mg BD (N=21)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Addominal Distention (Gastrointestinal disorders) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) — COVID-19 infection.
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT04618744/Prot_SAP_000.pdf